CLINICAL TRIAL: NCT03184181
Title: Application of Ultrasound-guided Electrolysis, Percutaneous Neuromodulation and Eccentric Exercise in Supraspinatus Tendinopathy
Brief Title: Application of Percutaneous Electrolysis, Percutaneous Neuromodulation and Eccentric Exercise
Acronym: MRH-EPTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Collaborators: Jorge Manuel Góngora Rodriguez (Unknown); Manuel Rodriguez Huguet (Unknown); Pablo Rodriguez Huguet (Unknown); Rocío Martín Valero (Unknown)
Responsible Party: Principal Investigator, Manuel Rodriguez Huguet, Degree Physiotherapy, University of Cadiz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 168/16
Record Dates: First submitted 2017-06-06; First posted 2017-06-12 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Supraspinatus Tendinitis
Keywords: tendinopathy; electrolysis; exercise; dry needling
MeSH Terms: conditions — Tendinopathy; Motor Activity

STUDY DESIGN:
Intervention Model Description: A specialist physician will be diagnosed the supraspinatus tendinopathy.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EPTE® group (Experimental): The intervention for this group consisted of Therapeutic Percutaneous Electrolysis (EPTE®). Patient received EPTE® once week for four weeks associated with eccentric exercises device at home.
  Interventions: Other: EPTE® group
- Dry needling group (Active Comparator): The intervention for this group consisted of dry needling in trigger points associated with eccentric exercises device at home. Patient received 3 sessions of dry needling a week for four weeks.
  Interventions: Other: Dry needling group

INTERVENTIONS:
Other: EPTE® group — Therapeutic Percutaneous Electrolysis once week for four weeks associated with eccentric exercises devices at home.
  Other Names: EPTE + EXER
  Arms: EPTE® group
Other: Dry needling group — The intervention for this group consisted of dry needling in trigger points associated with eccentric exercises devices at home.
  Other Names: DN + EXER
  Arms: Dry needling group

SUMMARY:
The supraspinatus muscle tendinopathy show a big impact, however, there is a lack of awareness about the options of the physiotherapist treatment. It is necessary to do studies about effectiveness of therapeutic percutaneous electrolysis (EPTE®). This technique enables treatment of the tendinopathies and the broken muscle fibrilare. It is base on the application of galvanic current through a acupuncture needle. To analyze the effectiveness of therapeutic percutaneous electrolysis (EPTE®) in the treatment of supraspinatus muscle tendinopathy. Single center randomized controlled trial, parallel treatment design. A specialist physician will be diagnosed the supraspinatus muscle tendinopathy. Participants will be randomly assigned to receive treatmen for 4 weeks: EPTE® associated with eccentric exercises or dry needling with the same eccentric exercises. Both interventions were performed under ultrasound guidance with a portable ultrasound (General Electric LogicE). Data will be collected by a blinded evaluator.

DETAILED DESCRIPTION:
Eccentric exercises of the supraspinatus muscle were performed in 3 sets of 10 repetitions. Participants were asked to perform the exercise program on an individual basis twice every day for 4 weeks. The eccentric program consisted of 3 exercises, focusing on the supraspinatus, infraspinatus, and scapular muscles. Participants were asked to do a normal abduction (concentric phase) and a slow return to the initial position (eccentric phase) included first the concentric phase, and the eccentric phase was slowly conducted. The exercise program was taught by a physiotherapist in the first session and monitored in the subsequent sessions.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with supraspinatus tendinopathies that do not improve with conventional physiotherapy or pharmacological therapy protocols.
* Subjects who are in an active state of pain, who present painful symptoms in a sensitive and painful area of the tendon of insertion of the supraspinatus muscle in the humerus.

Exclusion Criteria:

* Individuals who have received surgery intervention in the same shoulder, or have suffered fractures or dislocations in the same shoulder.
* Individuals have received the proposed treatment in one month´s period previously.
* Individuals who suffering from cervical radiculopathies, fibromialgia síndrome, cardiac patients with pacemakers, cancer, infectious processes, or generalized lymphedema.
* Pregnant women can not receive this treatment intervention.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
The intensity of shoulder pain | Baseline
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of shoulder pain, and the worst and lowest level of pain experienced in the preceding week in the shoulder area. The minimal clinically important difference (MCID) for the NPRS in patients with shoulder pain was 1.1 points (Mintken, Glynn, and Cleland 2009).

SECONDARY OUTCOMES:
The intensity of shoulder pain | Four weeks
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of shoulder pain, and the worst and lowest level of pain experienced in the preceding week in the shoulder area. The minimal clinically important difference (MCID) for the NPRS in patients with shoulder pain was 1.1 points (Mintken, Glynn, and Cleland 2009).
The intensity of shoulder pain | Eight weeks
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of shoulder pain, and the worst and lowest level of pain experienced in the preceding week in the shoulder area. The minimal clinically important difference (MCID) for the NPRS in patients with shoulder pain was 1.1 points (Mintken, Glynn, and Cleland 2009).
The intensity of shoulder pain | One year
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of shoulder pain, and the worst and lowest level of pain experienced in the preceding week in the shoulder area. The minimal clinically important difference (MCID) for the NPRS in patients with shoulder pain was 1.1 points (Mintken, Glynn, and Cleland 2009).
Active shoulder range of motion | Baseline, four weeks and one year.
  Measured by a two branches goniometer
Pressure pain thresholds in supraspinatus trigger points | Baseline, four weeks and one year.
  Pressure pain thresholds (PPTs) will be measured with a pressure algometer (Baseline, Pain TestTM, Wagner Instruments). The clinimetric properties of this instrument have been evaluated previously. The PPT will the point at which pressure elicited pain and will presented as kilograms per square centimeter. All measurements will be conducted by the same well-trained physician.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Manuel, BSc, Principal Investigator — University of Cadiz
Locations (1):
- Policlínica Santa María, Cadiz, Cádiz, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arias-Buria JL, Truyols-Dominguez S, Valero-Alcaide R, Salom-Moreno J, Atin-Arratibel MA, Fernandez-de-Las-Penas C. Ultrasound-Guided Percutaneous Electrolysis and Eccentric Exercises for Subacromial Pain Syndrome: A Randomized Clinical Trial. Evid Based Complement Alternat Med. 2015;2015:315219. doi: 10.1155/2015/315219. Epub 2015 Nov 15. PMID 26649058
- [Background] Mintken PE, Glynn P, Cleland JA. Psychometric properties of the shortened disabilities of the Arm, Shoulder, and Hand Questionnaire (QuickDASH) and Numeric Pain Rating Scale in patients with shoulder pain. J Shoulder Elbow Surg. 2009 Nov-Dec;18(6):920-6. doi: 10.1016/j.jse.2008.12.015. Epub 2009 Mar 17. PMID 19297202